CLINICAL TRIAL: NCT04811001
Title: A Randomised Non-comparative, Phase II Study Investigating the Best Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI) Sequence in Advanced or Metastatic Non Small-Cell Lung Cancer (NSCLC) Harboring EGFR Mutations
Brief Title: Best EGFR-TKI Sequence in NSCLC Harboring EGFR Mutations
Acronym: CAPLAND
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Ricerca Traslazionale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPLAND
Record Dates: First submitted 2021-01-28; First posted 2021-03-23 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: NSCLC
MeSH Terms: interventions — osimertinib; dacomitinib

STUDY DESIGN:
Intervention Model Description: Randomized, non-comparative study investigating two EGFR-TKI sequences
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Osimertinib->Dacomitinib) (Experimental): Osimertinib 80 mg/day until progression, unacceptable toxicity or patient refusal.
  At treatment discontinuation patients maintaining the original EGFR mutation will switch to Dacomitinib 45 mg/day until progression, unacceptable toxicity or patient refusal.
  Interventions: Drug: Osimertinib; Drug: Dacomitinib
- Arm B (Dacomitinib->Osimertinib) (Experimental): Dacomitinib 45 mg/day until progression, unacceptable toxicity or patient refusal.
  At treatment discontinuation, patients harboring the EGFR-T790M will receive Osimertinib 80 mg/day until progression, unacceptable toxicity or patient refusal.
  Interventions: Drug: Osimertinib; Drug: Dacomitinib

INTERVENTIONS:
Drug: Osimertinib — TAGRISSO 40 mg film-coated tablets TAGRISSO 80 mg film-coated tablets
  Other Names: Tagrisso
Drug: Dacomitinib — Vizimpro 15 mg film-coated tablets Vizimpro 30 mg film-coated tablets Vizimpro 45 mg film-coated tablets
  Other Names: Vizimpro

SUMMARY:
The best drug sequencing of dacomitinib or osimertinib in patients with advanced or metastatic Epidermal Growth Factor Receptor (EGFR) mutation positive non-small-cell lung cancer (NSCLC) has not yet been determined. The study enables investigation of the efficacy of dacomitinib followed by or subsequent to osimertinib osimertinib in patients with classical or uncommon activating EGFR mutations. Efficacy of dacomitinib will be defined in patients with asymptomatic or controlled brain metastases, special population eligible in this clinical trial.

DETAILED DESCRIPTION:
NSCLC remains the leading cause of cancer death in Western Countries. Lung adenocarcinoma has been extensively investigated and during the last 10 years several molecular events, including mutations, gene copy number alterations and translocations have been discovered, leading to a dramatic change in patient treatment. This is the case of EGFR mutant NSCLC in which drugs targeting the EGFR, such as gefitinib, erlotinib or afatinib, have demonstrated superiority versus standard chemotherapy. Osimertinib, (AZD9291, Tagrisso, AstraZeneca) is a third-generation EGFRTKI which irreversibly and specifically targets both sensitizing and the resistant T790M-mutated EGFRs. It has shown greater efficacy against EGFR T790M mutation than the standard platinum plus pemetrexed therapy and was thus recently fully approved by the FDA for metastatic EGFR T790M-positive NSCLC1. More recently, the large phase III FLAURA study, comparing osimertinib versus the first-generation EGFR-TKIs gefitinib or erlotinib, demonstrated the superiority of osimertinib in terms of progression-free survival (PFS; median PFS 18.9 months versus 10.2 months; HR: 0.46; p<0.0001)2. Based on this result, in October 2017, the FDA has granted Breakthrough Therapy Designation (BTD) for osimertinib for the first-line treatment of patients with metastatic EGFR mutation-positive NSCLC. In addition, the FLAURA trial clearly established the superiority of osimertinib even in special populations, including individuals with brain metastases. Due to these results, international consensus confirms osimertinib to be the standard of care as first-line therapy for NSCLC patients with EGFR M+ and as second-line therapy in patients with clinically relevant progression and confirmed T790M+. Dacomitinib (PF-00299804, Pfizer) is a second-generation, irreversible EGFRTKI, that has shown efficacy in NSCLC patients with EGFR mutations. Preclinical data showed that the drug is more potent than first-generation EGFR-TKIs, thus leading to comparative studies. The phase III ARCHER 1050 trial compared first-line dacomitinib versus gefitinib in patients with EGFR Del19 or L858R mutation-positive NSCLC. The trial met its primary endpoint, demonstrating a PFS improvement in favor of dacomitinib, (median PFS 14.7 months versus 9.2 months; HR: 0.59; p<0.0001) and, most importantly, it significantly prolonged OS (median OS 34.1 months versus 26.8 months; HR: 0.76; p=0.048). The most frequent adverse events (AEs) with dacomitinib were diarrhea, skin rash and stomatitis, requiring dose reduction in more than 60% of patients3. Importantly, patients with brain metastases were excluded precluding any conclusion on dacomitinib efficacy in this clinically relevant subgroup. Even with such limitations, indirect comparison with FLAURA showed that PFS was similar to that obtained with osimertinib, particularly in the Asian population, raising the question on the optimal sequencing of drugs. Data from different phase III studies suggested that median PFS with first- or second-generation EGFR-TKIs followed by osimertinib could be superior to the current standard of care, which is osimertinib followed by platinum-based chemotherapy. An important consideration is that only a fraction of patients receiving first- or second-generation EGFR-TKIs are eligible for osimertinib, because EGFR-T790M mutation occurs in up to 50% of cases. Therefore, at present, platinum-based chemotherapy is the only available option for EGFR-T790M negative patients. This algorithm is supported by the lack of efficacy of immunotherapy in presence of EGFR mutations, even if no study so far has been specifically conducted in patients progressing to first-line EGFRTKIs.

Optimised EGFR TKI sequencing might be the most critical determinant of OS in patients with activating EGFR mutations. Data on OS will help to understand the best sequence for each individual patient. Based on these premises, there is a strong rationale for conducting a trial exploring the best EGFR-TKI sequencing (i.e., that to achieve optimal clinical outcomes) in advanced or metastatic NSCLC individuals with EGFR mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. Male or female patient aged ≥18 years;
3. Histologically/cytologically confirmed diagnosis of stage IIIB/IV NSCLC with evidence of activating EGFR mutations including exon 19 deletion, exon 21 L858R or other activating/sensitizing EGFR mutations such as exon 21 L861Q, exon 18 G719S, G719A, G719C, exon 20 S768I and V769L; co-occurrence of de novo T790M is not an exclusion criterion; EGFR status assessed in circulating DNA is allowed;
4. Patients eligible and candidate to receive osimertinib as first- or second-line treatment according to clinical practice and study design, as decided by Investigator regardless study participation;
5. Patients with brain metastases are allowed provided they are asymptomatic and stable (i.e. without evidence of progression by imaging for at least two weeks prior to the first dose of trial treatment and without deterioration of any neurologic symptoms);
6. No evidence of concomitant drivers including KRAS mutations, HER2 mutations, ALK or ROS1 rearrangements, MET mutations, BRAF mutations;
7. No previous EGFR-TKI therapy; Previous palliative radiotherapy or surgery allowed. Prior brain radiotherapy and Stereotactic Radiosurgery (SRS) are allowed. Previous neo/adjuvant chemotherapy is allowed as long as therapy was completed at least 6 months before diagnosis of advanced or metastatic NSCLC;
8. At least one radiological measurable disease according to RECIST criteria version 1.1;
9. Performance status 0-1 (ECOG PS);
10. Patient compliance to trial procedures;
11. Adequate bone marrow function (ANC ≥ 1.5x109/L, platelets ≥100x109/L, haemoglobin >9 g/dl);
12. Adequate liver function (AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN, bilirubin < grade 2, transaminases no more than 3xULN/<5xULN in presence of liver metastases);
13. Normal level of alkaline phosphatase, and creatinine;
14. Female patients should be using adequate contraceptive measures, should not be breastfeeding, until 12 months after the last dose, and must have a negative pregnancy test (serum or urine) prior to first dose of study drug (within 72 hours); or female patients must have an evidence of non-childbearing potential by fulfilling one of the following criteria at screening:

    * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
    * Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the institution. Documentation of irreversible surgical by hysterectomy, bilateraloophorectomy, or bilateral salpingectomy but not tubal ligation.
15. Male patients should be willing to use barrier contraception, i.e. condoms;
16. No significant comorbidity that according to the investigator would hamper the participation on the trial;

Exclusion Criteria:

1. Previous therapy with any EGFR-TKI;
2. Previous systemic anti-cancer therapy for advanced/metastatic NSCLC including chemotherapy, biologic therapy, immunotherapy, or any investigational drug;
3. Absence of measurable lesions;
4. Concomitant radiotherapy or chemotherapy;
5. Symptomatic or immediately requiring therapy brain metastases or carcinomatous meningitis. Subjects with asymptomatic and stable or treated brain metastases may participate;
6. Diagnosis of any other malignancy during the last 3 years, except for in situ carcinoma of cervix uteri and squamous cell carcinoma of the skin;
7. History of extensive disseminated/bilateral or known presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis and pulmonary fibrosis (but not history of prior radiation pneumonitis);
8. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses; or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV);
9. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of the study drugs;
10. Any of the following cardiac criteria:

    * Mean resting corrected QT interval (QTc) >470 msec, obtained from 3 ECGs using local clinic ECG machine-derived QTcF value;
    * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG, e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250 msec or history of episodes of bradycardia (<50 BPM);
    * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval;
    * Abnormal cardiac function: LVEF < 50% (assessed by MUGA or ECHO)
11. Pregnancy or lactating female;
12. Other serious illness or medical condition potentially interfering with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 2 years since last patient enrolled
  OS defined as the time from randomization to the date of death due to any cause, or to the date of censoring at the last time the subject was known to be alive

SECONDARY OUTCOMES:
Progresison Free Survival (PFS1) | Up to 2 years since last patient enrolled
  PFS1 defined the time from randomization to disease progression or death from any cause
Progresison Free Survival (PFS2) | Up to 2 years since last patient enrolled
  PFS2 defined the time from second line treatment start to disease progression or death from any cause
Response Rate (RR) | At 1 year and 2 years
  RR defined as the percentage of patients whose cancer shrinks or disappears after study treatment
Adverse Events | During the trial, untill 2 years
  Incidence of Adverse Events in patients treated with osimertinib followed by dacomitinib or with the opposite sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Morabito, MD, Principal Investigator — Istituto Nazionale Tumori IRCCS Fondazione Pascale
Locations (20):
- Italy (20):
  - Istituto Toscano Tumori Ospedale San Donato, Arezzo, AR
  - IRCCS Istituto Tumori "Giovanni Paolo II", Bari, BA
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.), Meldola, FC
  - ca Azienda OspedalieroUniversitaria Caregg, Florence, FI
  - IRCCS AOU San Martino IST - Istituto Nazionale per la Ricerca sul Cancro, Genova, GE
  - Ospedale Versilia, Lido di Camaiore, LU
  - Ospedale San Luca, Lucca, LU
  - AOU - Policlinico di Modena, Modena, MO
  - Azienda Ospedaliera Universitaria Paolo Giaccone, Palermo, PA
  - Casa di Cura La Maddalena, Palermo, PA
  - Istituto Oncologico Veneto, Padua, PD
  - Centro di Riferimento Oncologico di Basilicata, Rionero in Vulture, PZ
  - RCCS- Arcispedale Santa Maria Nuova, Reggio Emilia, RE
  - Istituto Nazionale Tumori "Regina Elena", Roma, RM
  - Ospedale Civile SS. Annunziata, Sassari, SS
  - Azienda Ospedaliera S. Maria di Terni, Terni, TR
  - A.O. Busto Arsizio P.O. Saronno, Saronno, VA
  - ASST Sette Laghi, Varese, VA
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - A.O.U. "Maggiore della Carità, Novara